CLINICAL TRIAL: NCT00917891
Title: A Double-blind, Randomized, Placebo-Controlled Phase I/II Study to Evaluate the Safety and Acceptability of Dapivirine Gel 4759, 0.05%, 2.5g, a Vaginal Microbicide, Conducted Using Daily Monitored Adherence in Healthy, HIV-Negative Women.
Brief Title: An Expanded Safety Study of Dapivirine Gel 4759 in Africa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IPM 014A
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome
Keywords: HIV Infections; Acquired Immunodeficiency Syndrome; Healthy; HIV seronegativity
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Dapivirine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vehicle placebo gel (Placebo Comparator)
  Interventions: Drug: placebo
- dapivirine gel (Experimental)
  Interventions: Drug: dapivirine

INTERVENTIONS:
Drug: dapivirine — dosage form: vaginal gel
  dosage: 1.25mg dapivirine/day
  frequency: once daily
  duration: 6 weeks
  Arms: dapivirine gel
Drug: placebo — dosage form: vaginal gel
  frequency: once daily
  duration: 6 weeks
  Arms: vehicle placebo gel

SUMMARY:
The purpose of this study is to determine whether dapivirine gel 4759 is safe for daily use by healthy women in Kenya, Malawi, Rwanda, South Africa and Tanzania.

DETAILED DESCRIPTION:
To reduce the influence of adherence as a factor in the interpretation of efficacy results, IPM is considering using a DOT (Directly Observed Therapy) based method for vaginal microbicide gel delivery in a future Phase III study. IPM has denoted this DOT based method as Daily Monitored Adherence (DMA). IPM014A is a Phase I/II study designed: (1) to assess and compare the safety of a once daily application of Dapivirine Gel 4759, 0.05% 2.5g and a matching vehicle placebo gel; (2) to assess the acceptability of a once daily application of Dapivirine gel 4759, 0.05% 2.5g and a matching vehicle placebo gel; and (3) to assess the feasibility of utilizing the DMA method for a large-scale phase III efficacy study.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 to 40 years of age inclusive who can give written informed consent
2. Available for all visits and consent to follow all procedures scheduled for the study
3. Agree to daily application of gel and monitoring as per Daily Monitored Adherence (DMA) method
4. Healthy and self-reported sexually active
5. HIV-negative as determined by a HIV rapid test at time of enrollment
6. On a stable form of contraception and willing to continue on this stable method of contraception, OR, Have undergone surgical sterilisation at least 3 months prior to enrollment
7. In the absence of the use of exogenous hormone(s), have a self-reported regular menstrual cycle defined as having a minimum of 21 days and a maximum of 36 days between menses
8. Upon pelvic/speculum examination and colposcopy at the time of enrollment, the cervix and vagina appear normal as determined by the investigator
9. Asymptomatic for genital infections at the time of enrollment
10. Willing to refrain from use of vaginal products or objects within 14 days prior to enrollment and for the duration of the study
11. Willing to answer acceptability and adherence questionnaires throughout the study
12. Willing to refrain from participation in any other research study for the duration of this study
13. Willing to provide adequate locator information for study retention purposes and be reachable per local standard procedures

Exclusion Criteria:

1. Currently pregnant or last pregnancy outcome within 3 months prior to enrolment
2. Currently breast-feeding
3. Participated in any other research study within 60 days prior to screening
4. Previously participated in any HIV vaccine study
5. Untreated urogenital infections (either symptomatic or asymptomatic) within 2 weeks prior to enrollment
6. Presence of abnormal physical finding on the vulva, vaginal walls or cervix during pelvic/speculum examination and/or colposcopy
7. History of significant urogenital or uterine prolapse, undiagnosed vaginal bleeding, urethral obstruction
8. Pap smear result at screening that requires cryotherapy, biopsy, treatment (other than for infection), or further evaluation
9. Any Grade 2, 3 or 4 baseline haematology, chemistry or urinalysis laboratory abnormality according to the DAIDS Table for Grading Adverse Experiences
10. Unexplained, undiagnosed abnormal bleeding per vagina, bleeding per vagina during or following vaginal intercourse, or gynaecologic surgery within 90 days prior to enrollment
11. Any history of anaphylaxis or severe allergy resulting in angioedema; or a history of sensitivity/allergy to latex
12. Any serious acute, chronic or progressive disease
13. Any condition(s) that, in the opinion of the investigator, might interfere with adherence to study requirements or evaluation of the study objectives

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 280 (Actual)
Dates: Start 2009-11; Primary Completion 2011-01 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Gynaecological examinations, including pelvic/speculum examination and colposcopy, and laboratory STI testing. | Week 0, 1, 2, 4, 6 & 10
Safety laboratory tests | enrollment & last day of gel use
Adverse event/serious adverse event reports | throughout study

SECONDARY OUTCOMES:
Questionnaires concerning acceptability and adherence to daily use of vaginal gel. | Week 0, 2, 6 & 10
Documentation of adherence to the DMA method including the Applicator Collection Checklist, focus groups and male interviews. | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Dr Annalene Nel, Study Director — Beijing Immupeutics Medicine Technology Limited
Locations (10):
- Kenya Medical Research Institute, Kisumu, Kenya
- Johns Hopkins Project, College of Medicine, Blantyre, Malawi
- Projet Ubuzima, Kigali, Rwanda
- South Africa (6):
  - Be Part Clinic, Mbekweni, Paarl, Eastern Cape
  - Qhakaza Mbokodo, Ladysmith, KwaZulu-Natal
  - Prevention for HIV and AIDS Project, Pinetown, KwaZulu-Natal
  - Ndlela HIV Research and Clinical Tirals Unit, Agincourt, Mpumalanga
  - Madibeng Centre for Research, Brits, North West
  - Desmond Tutu HIV Foundation, Nyanga, Cape Town, Western Cape
- Kilimanjaro Christian Medical Centre, Moshi, Tanzania